CLINICAL TRIAL: NCT00827697
Title: A Validation Study of the Gen-Probe APTIMA Combo2 (AC2) for Detecting Chlamydia Trachomatis and Neisseria Gonorrhoeae in Rectal Samples.
Brief Title: A Validation Study for Detecting Chlamydia and Gonorrhea in Rectal Samples
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sharon Hillier, Richard Sweet Professor of Reproductive Infectious Disease, University of Pittsburgh
Other Study IDs: PRO08120504; UM1AI068633 (NIH); 5UM1AI106707 (NIH)
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Gonorrhea; Chlamydia
Keywords: Gonorrhea; Chlamydia; Rectal
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Gen-Probe APTIMA Combo2 (AC2) — Laboratory Test

SUMMARY:
Our hypothesis is that nucleic acid amplification testing (NAAT) with the APTIMA Combo2 (AC2) will have greater sensitivity than culture in detecting Neisseria gonorrhoeae in rectal samples. We also hypothesize that AC2 will be equivalent to NAAT with the Becton Dickinson ProbeTec in detecting Chlamydia trachomatis and Neisseria gonorrhoeae in rectal samples.

DETAILED DESCRIPTION:
This research is being done to compare the results of tests for diagnosing sexually transmitted infections (STI) from rectal samples. Specifically, this study will test for gonorrhea and Chlamydia from rectal samples and compare the results between standard culture and newer technology (nucleic acid amplification testing otherwise know as "NAAT") used to detect these infections. Gonorrhea and Chlamydia are STIs (infections you get from having sex with someone who is infected). Infections in the rectum may cause symptoms such as rectal discharge, itching and/or pain or may be asymptomatic (no symptoms present). Since these infections are sexually transmitted, it is important to have accurate tests to diagnose and treat these infections to prevent them from being passed onto a sexual partner.

NAAT has not been Food and Drug Administration (FDA) approved for use in diagnosing these infections in the rectum. The tests are approved to detect these infections from other sites (cervix and urine) and investigators believe that these tests will be very accurate in detecting these infections in the rectum as well. This study will validate the use of NAAT in rectal samples so that this technology can be used in our research laboratory for future studies that involve testing for STIs from the rectum.

There are times when people have signs of inflammation in the rectum (known as proctitis) and an infection or cause is not able to be identified. Investigators believe that this new technology (NAAT) may be able to find reasons (different bacteria) for infection that were not able to be identified with older testing methods. By participating in this study, one of the rectal swabs will also be tested for additional bacteria (called Mycoplasma and Trichomonas). Both of these organisms are sexually transmitted and may be important organisms in the cause of proctitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 and older
2. Women or men who have a history of engaging in receptive anal intercourse
3. Willing to provide written informed consent for participation in this study

Exclusion Criteria:

1. Use of oral antibiotics in the past 7 days
2. Use of rectal douche or other rectal product in the past 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women (n=175) and men who have sex with men (n=224) with a lifetime history of anal intercourse by self-report
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of AC2 in detecting Neisseria gonorrhoeae in rectal samples | Visit 1
  Sensitivity and specificity of AC2 to ProbeTec and culture in detecting Neisseria gonorrhoeae in rectal samples
Sensitivity and specificity of AC2 in detecting Chlamydia trachomatis in rectal samples | Visit 1
  Compare the sensitivity and specificity of the AC2 to ProbeTec and as necessary, for discrepant results, to APTIMA CT assay in detecting Chlamydia trachomatis in rectal sample

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Pittsburgh AIDS Center for Treatment (PACT), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No